CLINICAL TRIAL: NCT00000977
Title: Active Immunization of Asymptomatic, HIV-Infected Individuals With Recombinant GP160 HIV-1 Antigen: A Phase I/II Study of Immunogenicity and Toxicity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Protein Sciences Corporation (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 137; 11112 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV Seropositivity; HIV-1; Drug Evaluation; AIDS Vaccines; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections; HIV Seropositivity | interventions — VaxSyn HIV-1 (gp160) vaccine

INTERVENTIONS:
Biological: gp160 Vaccine (MicroGeneSys)

SUMMARY:
To determine the minimal effective (immunogenic) dose of vaccine in asymptomatic HIV-1 seropositive individuals with > 400 cells/mm3 (CD4). To determine the dose-response to a 4 fold escalation of the immunizing dose. To describe both cellular and humoral immune responses to HIV-1 in the immunized individuals. To describe the effects of this immunization on general immunological, virological and clinical parameters. To evaluate the safety of injecting recombinant gp160 in this population. To evaluate the extent of variability between different lots of gp160 (arms C1 and C2). It might be possible to increase immune responses or to induce new types of immune responses to HIV in some infected individuals by means of a vaccine, which could result in an immunological, virological or clinical benefit.

DETAILED DESCRIPTION:
It might be possible to increase immune responses or to induce new types of immune responses to HIV in some infected individuals by means of a vaccine, which could result in an immunological, virological or clinical benefit.

ORIGINAL DESIGN: Patients are randomized to one of five groups to receive, intramuscularly, one of four dosages of gp160 or hepatitis B vaccine as a control. Treatments are given at 0, 1, 3, 6, 9, and 12 months and patients are followed for up to 2 years. Patients in any of the 5 groups will have the option of switching to another dosage group if an interim analysis at 6 months shows significant differences in patient response. AMENDED: 10/23/90 52 eligible patients are randomized to one of 6 study groups. Five groups of 8 individuals receive one of 4 dosage levels of gp160 (Groups A, B, C1, C2, and D), and 12 patients receive a single dosage level of hepatitis B vaccine as a control (Group E). Per 2/19/92 amendment, patients may elect to continue receiving vaccine beyond 12 months, with the doses given either every 3 months or every 6 months.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Acute use (< 14 days) of acyclovir for Herpes simplex virus infection or ketoconazole for symptomatic Candida infections.

An additional group of up to 20 patients may be added to the study. Patients from ACTG 148 with a repeatedly negative delayed-type hypersensitivity (DTH) reaction who have reached their third dose of ID gp160 at 32 mcg and have failed to develop new proliferative response have the option, after a 2-month interval, to enter this protocol.

* They must meet inclusion and exclusion criteria that apply to this protocol.
* Patients with CD4 counts of 400 - 500 cells/mm3 must be informed of the recommended zidovudine (AZT) therapy and sign an informed consent statement declining AZT therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Fever of > 100 degrees F persisting for > 15 days in a 30-day interval without definable cause.
* Recurrent oral candidiasis.
* Multidermatomal herpes zoster.
* Biopsy-proven hairy leukoplakia.
* Fatigue/malaise of > 1 month duration that interferes with normal activities.
* Evidence of clinically significant central nervous system dysfunction as assessed by neurological exam.
* Involuntary weight loss > 10 lbs or 10 percent of normal weight in a 6 month interval.
* Diarrhea (> 3 stools/day) for more than 30 days without definable cause.

Concurrent Medication:

Excluded:

* Antiretroviral agents of proven or potential efficacy or any potential immunoenhancing or immunosuppressive drugs.

Patients with the following are excluded:

* Known hypersensitivity to insect cells or baculovirus.
* Abnormal chest x-ray taken within 3 months of study entry.
* Systemic symptoms thought to be due to HIV infection (other than lymphadenopathy). Evidence of clinically significant central nervous system dysfunction as assessed by neurological exam.
* Unwilling or unable to give written informed consent.

Prior Medication:

Excluded within 90 days of study entry:

* Zidovudine (AZT), didanosine (ddI), or any potential antiretroviral or immunomodulating agents.

Active substance abuse (either continuing daily alcohol abuse or intravenous drug use).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52
Dates: Study Completion 1993-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valentine F, Study Chair
Locations (2):
- United States (2):
  - Stanford CRS, Palo Alto, California
  - NY Univ. HIV/AIDS CRS, New York, New York

REFERENCES:
- [Background] Katzenstein DA, Kundu S, Spritzler J, Smoller BR, Haszlett P, Valentine F, Merigan TC. Delayed-type hypersensitivity to recombinant HIV envelope glycoprotein (rgp160) after immunization with homologous antigen. J Acquir Immune Defic Syndr. 1999 Dec 1;22(4):341-7. doi: 10.1097/00126334-199912010-00004. PMID 10634195
- [Background] Kundu SK, Katzenstein D, Valentine FT, Spino C, Efron B, Merigan TC. Effect of therapeutic immunization with recombinant gp160 HIV-1 vaccine on HIV-1 proviral DNA and plasma RNA: relationship to cellular immune responses. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Aug 1;15(4):269-74. doi: 10.1097/00042560-199708010-00004. PMID 9292585
- [Background] Valentine F, et al. A randomized, controlled study of immunogenicity of rgp160 vaccine in HIV-infected subjects. Int Conf AIDS. 1992 Jul 19-24;8(1):Tu39 (abstract no TuB 0561)
- [Background] Valentine FT, Kundu S, Haslett PA, Katzenstein D, Beckett L, Spino C, Borucki M, Vasquez M, Smith G, Korvick J, Kagan J, Merigan TC. A randomized, placebo-controlled study of the immunogenicity of human immunodeficiency virus (HIV) rgp160 vaccine in HIV-infected subjects with > or = 400/mm3 CD4 T lymphocytes (AIDS Clinical Trials Group Protocol 137). J Infect Dis. 1996 Jun;173(6):1336-46. doi: 10.1093/infdis/173.6.1336. PMID 8648205
- [Background] Kundu SK, Katzenstein D, Moses LE, Merigan TC. Enhancement of human immunodeficiency virus (HIV)-specific CD4+ and CD8+ cytotoxic T-lymphocyte activities in HIV-infected asymptomatic patients given recombinant gp160 vaccine. Proc Natl Acad Sci U S A. 1992 Dec 1;89(23):11204-8. doi: 10.1073/pnas.89.23.11204. PMID 1360665